CLINICAL TRIAL: NCT01850810
Title: Evaluation of a Nutritional Product for People With Type 2 Diabetes (T2DM)
Brief Title: Evaluation of a Nutritional Product for People With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BL17
Record Dates: First submitted 2013-05-06; First posted 2013-05-10 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Study Product (Experimental): 1 serving of a nutritional product for people with diabetes.
  Interventions: Other: Experimental Study Product
- Control Study Product (Placebo Comparator): 1 serving of control beverage.
  Interventions: Other: Control Study Product

INTERVENTIONS:
Other: Experimental Study Product
  Other Names: Oral nutritional supplement for people with Diabetes.
  Arms: Experimental Study Product
Other: Control Study Product
  Other Names: Water beverage.
  Arms: Control Study Product

SUMMARY:
The objective of this trial is to evaluate a nutritional product for people with Diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible for the study if they meet all of the following inclusion criteria:

  1. Diagnosis of Type 2 Diabetes.
  2. Age between 18 and 75 years.
  3. HbA1c > 6.0 but ≤ 8.5
  4. If female and of childbearing potential , subject is non-pregnant, non- lactating, at least 6 weeks postpartum and agrees to practice birth control throughout study duration.
  5. BMI is > 18.5 kg/m2 and < 40.0 kg/m2.
  6. Chronic medication dosage must be stable for at least two months prior to Screening Visit.
  7. Subject states that they are a habitual consumer of a morning meal.

Exclusion Criteria:

* Subjects will be excluded from the study if they meet any of the following criteria:

  1. Use of exogenous insulin or GLP-1 agonists for glucose control.
  2. Diagnosis of Type 1 diabetes.
  3. History of diabetic ketoacidosis.
  4. Current infection (requiring medication or hospitalization), has received corticosteroid treatment in the last 3 months, or has had surgery or received antibiotics in the last 3 weeks.
  5. Active malignancy.
  6. Significant cardiovascular event < 12 weeks prior to study entry.
  7. End stage organ failure or status post organ transplant.
  8. Active metabolic, hepatic, or gastrointestinal disease.
  9. Chronic, contagious, infectious disease.
  10. Currently taking herbals, dietary supplements, or medications (other than antihyperglycemic medications) that could profoundly affect blood glucose.
  11. History of fainting or other adverse reactions in response to blood collection.
  12. Clotting or bleeding disorders.
  13. Allergy or intolerance to study product ingredient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Hunger | Treatment Visit Week 1 and Treatment Visit Week 2
  An appetite questionnaire administered 0 to 300 minutes during each study visit.

SECONDARY OUTCOMES:
Fullness | Treatment Visit Week 1 and Treatment Visit Week 2
  An appetite questionnaire administered 0 to 300 minutes during each study visit.
Desire to Eat | Treatment Visit Week 1 and Treatment Visit Week 2
  An appetite questionnaire administered 0 to 300 minutes during each study visit.
Prospective Consumption | Treatment Visit Week 1 and Treatment Visit Week 2
  An appetite questionnaire administered 0 to 300 minutes during each study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Devitt-Maicher, PhD, Study Chair — Abbott Nutrition
Locations (2):
- United States (2):
  - Radiant Research, Chicago, Illinois
  - Radiant Research, Cincinnati, Ohio